CLINICAL TRIAL: NCT07075497
Title: Short Term Effects of Proprioceptive Neuromuscular Facilitation Combined With Neuromuscular Electrical Stimulation in Young Football Players: a Randomized Clinical Trial
Brief Title: Effects of Combining PNF With NMES in Young Football Players
Acronym: PNF+NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-97
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hamstring Flexibility; Hamstring Muscle Tightness
Keywords: hamstring flexibility; football; Propioceptive Neuromuscular Facilitation; Neuromuscular Electrical Stimulation; Sports Injury Prevention; Athletic Performance; Muscle Stretching; Hamstring Muscle Function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- contract-relax proprioceptive neuromuscular facilitation with sham NMES (crPNF + sham NMES) (Placebo Comparator): Participants sat in long-sitting with maximal knee extension and pelvic anteversion controlled by elastic straps over the pelvis and distal thigh. Two 5×5 cm self-adhesive electrodes were placed on the hamstrings: one two fingerbreadths below the gluteal fold (proximal) and one over the distal third of the muscle belly. Sham NMES delivered biphasic symmetric rectangular pulses (50 Hz, 250 µs) at the sensory threshold (minimal intensity eliciting only a slight tingling without visible muscle response). Each of three cycles comprised a 10 s maximal voluntary isometric hamstring contraction ("Squeeze…!") against the fixed table, immediately followed by a 30 s passive stretch to a moderate-strong but non-painful tension ("Stretch…!"). A primary researcher ensured consistent limb positioning and strap tension; a secondary researcher monitored timing and cued contractions by lightly supporting the heels.
  Interventions: Other: Sham Neuromuscular electrical stimulation (NMES); Other: Contract-Relax PNF (crPNF)
- Neuromuscular Electrical Stimulation (NMES + crPNF) (Experimental): Participants sat in long-sitting with maximal knee extension and pelvic anteversion controlled by elastic straps over the pelvis and distal thigh. Two 5×5 cm self-adhesive electrodes were placed on the hamstrings: one two fingerbreadths below the gluteal fold (proximal) and one over the distal third of the muscle belly. NMES delivered biphasic symmetric rectangular pulses (50 Hz, 250 µs) at each participant's maximal motor threshold without discomfort or pain; the resulting milliamperage was recorded for each leg and used during all contraction phases. Each of three cycles comprised a 10 s maximal voluntary isometric hamstring contraction ("Squeeze…!") with NMES applied at the recorded intensity, immediately followed by a 30 s passive stretch to a moderate-strong but non-painful tension ("Stretch…!"). A primary researcher ensured consistent limb positioning and strap tension; a secondary researcher monitored timing and cued contractions by lightly supporting the heels.
  Interventions: Other: Neuromuscular electrical stimulation (NMES); Other: Contract-Relax PNF (crPNF)

INTERVENTIONS:
Other: Neuromuscular electrical stimulation (NMES) — NMES is applied during each 10-second isometric hamstring contraction using an Enraf Nonius TensMed S82 stimulator delivering biphasic, symmetric rectangular pulses at 50 Hz with a 250 µs pulse width. Two 5 × 5 cm self-adhesive electrodes are placed on the hamstrings-one approximately two finger-breadths below the gluteal fold and the other over the distal third of the muscle belly. Stimulation intensity is individually titrated to each participant's maximal motor threshold-eliciting a strong, yet painless, contraction-and the exact milliamperage is recorded for each leg. Elastic straps over the pelvis and distal thigh maintain pelvic anteversion and knee extension. During each session, one researcher secures limb positioning while a second adjusts and logs NMES intensity and cues the timing of the 10 s contraction and ensuing 30 s passive stretch.
  Arms: Neuromuscular Electrical Stimulation (NMES + crPNF)
Other: Sham Neuromuscular electrical stimulation (NMES) — Sham NMES is delivered during each 10 s isometric hamstring contraction using an Enraf Nonius TensMed S82 stimulator with biphasic, symmetric rectangular pulses (50 Hz, 250 µs pulse width). Two 5 × 5 cm self-adhesive electrodes are placed on the hamstrings-one two finger-breadths below the gluteal fold and one over the distal third of the muscle belly. Intensity is individually set to the sensory threshold, defined as the minimal current producing a slight tingling without any visible muscle response; this milliamperage is recorded for each leg. Elastic straps over the pelvis and distal thigh maintain pelvic anteversion and full knee extension. During each session, one researcher secures limb positioning while a second adjusts and logs the NMES intensity and cues the 10 s contraction timing.
  Arms: contract-relax proprioceptive neuromuscular facilitation with sham NMES (crPNF + sham NMES)
Other: Contract-Relax PNF (crPNF) — The crPNF Group engages in an isolated contract-relax proprioceptive neuromuscular facilitation (crPNF) stretching protocol. Participants are positioned in a long sitting posture with maximum knee extension until they feel a moderate-strong stretch sensation, without pain. Each stretch lasts for 30 seconds, followed by a 10-second maximal voluntary isometric contraction of the hamstrings. Participants complete three cycles of stretch and contraction. One researcher maintains the stretch position while a second researcher controls the timing of the stretching and contractions.

SUMMARY:
Hamstring muscle injuries are common in sports like football and often lead to extended periods of inactivity. This study aims to compare the effects of two different stretching programs on hamstring flexibility, with a secondary focus on jumping performance in young football players. One group will perform a proprioceptive neuromuscular facilitation (PNF) stretching protocol combined with neuromuscular electrical stimulation (NMES), while the other group will follow the same PNF protocol with a placebo NMES.

DETAILED DESCRIPTION:
Hamstring strains are increasingly common in sports, particularly in football, where they are among the most frequent injuries. Stretching techniques such as proprioceptive neuromuscular facilitation (PNF) are commonly used to improve muscle flexibility and reduce injury risk. A specific variant, contract-relax PNF (crPNF), involves alternating passive stretching with voluntary muscle contractions. Recent approaches suggest that applying neuromuscular electrical stimulation (NMES) during the contraction phase of crPNF may further enhance its effectiveness.

This study aims to compare the short-term effects of two active stretching protocols on hamstring flexibility in young male football players. One group will perform crPNF with sham NMES, while the other will perform crPNF with NMES during the contraction phase. A secondary objective is to assess whether either protocol affects vertical jump performance, a key ability in football.

ELIGIBILITY:
Inclusion Criteria:

* Active football players who train at least 3 days a week.
* Ages between 10 and 18 years.

Exclusion Criteria:

* Are currently engaged in a structured hamstring-stretching programme.
* Present with acute low back pain.
* Have sustained a hamstring injury within the past 6 months.
* Have undergone spinal or abdominal surgery within the past 6 months.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-27 (Actual)

PRIMARY OUTCOMES:
The Popliteal Angle Test | Before and inmediately after the intervention
  The Popliteal Angle Test is validated for measuring hamstring extensibility. Participants are placed in the supine position. A researcher holds the hip at a 90° flexion and passively extends the knee until the participant feels a strong stretch without pain. The examiner records the knee extension degrees at that moment using an inclinometer. The test is repeated three times, and the average is obtained. A full knee extension corresponds to a value of 0 degrees, and a higher number of degrees indicates greater hamstring shortening.
The Sit & Reach Test | Before and inmediately after the intervention
  The Sit & Reach Test has high intra-examiner reliability and is validated for measuring hamstring extensibility. For its execution, participants are placed in a long sitting position with the soles of their feet against the base of the measurement box. Keeping their knees extended, they reach for the maximum possible distance in the box with their fingers. The test is repeated three times, and the average is obtained. Values are recorded in centimeters, where a greater distance indicates a higher degree of hamstring extensibility.

SECONDARY OUTCOMES:
The Counter Movement Jump | Before and inmediately after the intervention
  The Counter Movement Jump is validated and standardized in adolescents for measuring jumping ability. The instructions by Petrigna et al. are followed to perform the jump. The My Jump App is used, which has high reliability and validity for measuring vertical jump height in centimeters. A greater height indicates a greater jumping ability.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Lisón Párraga, Dr, Principal Investigator — Cardenal Herrera University
Locations (1):
- University Ceu Cardenal Herrera, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided